CLINICAL TRIAL: NCT00075491
Title: A Phase II Evaluation With Correlative Studies Of Fenretinide (NSC 374551-4HPR) As A Single Agent In The Treatment Of Adult Patients With Recurrent Glioblastoma Multiforme
Brief Title: Neoadjuvant and Adjuvant Fenretinide Compared With Adjuvant Fenretinide Alone in Treating Patients Who Are Undergoing Surgical Resection For Recurrent Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02566; ID02-701; R21CA097767 (NIH); CDR0000346722 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (fenretinide, surgery) (Experimental): Patients receive neoadjuvant oral fenretinide twice daily for 1 week and then undergo surgical resection.
  Interventions: Drug: fenretinide; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (surgery) (Active Comparator): Patients undergo surgical resection.
  Interventions: Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fenretinide — Given orally
  Other Names: fenretinimide; McN-R-1967
  Arms: Arm I (fenretinide, surgery)
Procedure: therapeutic conventional surgery — Undergo surgery
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well neoadjuvant and adjuvant fenretinide works compared to adjuvant fenretinide alone in treating patients who are undergoing surgical resection for recurrent glioblastoma multiforme. Chemotherapy drugs, such as fenretinide, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy before surgery may shrink the tumor so that it can be removed. Giving chemotherapy after surgery may kill any remaining tumor cells. It is not yet known whether neoadjuvant and adjuvant fenretinide is more effective than adjuvant fenretinide alone

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the efficacy of neoadjuvant and adjuvant fenretinide vs adjuvant fenretinide alone, in terms of 6-month progression-free survival, in patients with recurrent glioblastoma multiforme undergoing surgical resection II. Correlate the serum and glioma tissue pharmacology of this drug with clinical response in patients treated with these regimens.

III. Determine whether this drug induces apoptosis in glioma tissue in patients treated with these regimens.

IV. Correlate the apoptotic index with tissue and serum concentration and clinical response in patients treated with these regimens.

V. Compare radiological response, overall survival, and unexpected toxicity in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive neoadjuvant oral fenretinide twice daily for 1 week and then undergo surgical resection.

Arm II: Patients undergo surgical resection.

Beginning two weeks after surgery, all patients receive adjuvant oral fenretinide twice daily on weeks 1 and 4. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 21-46 patients (10-23 per treatment arm) will be accrued for this study within 7-46 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme after initial tumor resection
* Radiologically evident recurrent tumor after prior radiotherapy OR after treatment for no more than 2 prior relapses

  * Enhancing or nonenhancing recurrent disease by MRI
* No progressive symptoms requiring urgent surgery
* Performance status - Karnofsky 70-100%
* More than 8 weeks
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* PT/PTT no greater than upper limit of normal
* SGPT no greater than 2.5 times normal
* Alkaline phosphatase no greater than 2.5 times normal
* Bilirubin less than 1.5 mg/dL
* BUN no greater than 1.5 times normal
* Creatinine no greater than 1.5 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 2 months after study participation
* Amylase and lipase normal
* No active infection
* No other disease that would obscure toxicity or dangerously alter drug metabolism
* No other concurrent serious medical illness
* Not at risk from any study treatment delays
* Able to swallow fenretinide capsules
* Recovered from all prior chemotherapy
* Approximately 2 weeks since prior vincristine
* Approximately 6 weeks since prior nitrosoureas
* Approximately 3 weeks since prior procarbazine
* See Disease Characteristics
* At least 2 weeks since prior radiotherapy
* See Disease Characteristics
* At least 1 week since prior vitamin A
* At least 1 week since prior isotretinoin (Accutane®)
* No concurrent vitamin A during and for 2 weeks after study participation
* No concurrent antioxidants (e.g., ascorbic acid or vitamin E)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 6 months
Plasma and tissue concentrations of fenretinide and its metabolite, 4-MPR using high-performance liquid chromatography (HPLC) assay | At baseline, and at 1, 7, 14, and 21 days
Tumor apoptotic index after fenretinide treatment by immunohistochemistry | At the time of surgery
Correlation between tumor apoptotic index with serum and tissue fenretinide levels | At the time of surgery
Correlation of time to progression with drug levels and apoptotic index | Up to 2 years

SECONDARY OUTCOMES:
Fenretinide effects on retinol, RBP, retinoid receptor levels and IGF-1 | Up to 21 days (course 1 and 4)
Fenretinide activity using magnetic resonance spectroscopy (MRS) | At the time of surgery
Radiological response | Up to 2 years
Overall survival | Up to 2 years
Unexpected toxicity associated with fenretinide as assessed by CTC version 3.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vinay K. Puduvalli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States